CLINICAL TRIAL: NCT02990871
Title: Efficacy of an Early Rehabilitation on Decannulation Time of Patients With Severe Acquired Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Other Study IDs: tracheostomy_01
Record Dates: First submitted 2016-09-29; First posted 2016-12-13 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Brain Injury; Tracheostomy; Neurological Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- early rehabilitation: Patients started rehabilitative treatment during ICU hospitalization
  Interventions: Other: early neurological rehabilitation
- no-early rehabilitation: Patients started rehabilitative treatment after admission in Neuro-rehabilitation department
  Interventions: Other: no-early neurological rehabilitation

INTERVENTIONS:
Other: early neurological rehabilitation — start of neurological rehabilitation between 3rd and 15th day after ABI
  Groups: early rehabilitation
Other: no-early neurological rehabilitation — start of neurological rehabilitation between 20th and 90th day after ABI
  Groups: no-early rehabilitation

SUMMARY:
All the patients hospitalized in the neuro-rehabilitation after a severe acquired brain injury carrying a tracheal cannula will be retrospectively analyzed. Patients coming from emergency department started a rehabilitative treatment during their hospitalization in ICU. Patients transferred from an external ICU started the rehabilitation in neurorehabilitation department. Aim of the study is to evaluate if an early rehabilitation, started since the acute stage of the damage, is able to reduce the decannulation time in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* presence of a tracheostomy at admission in NRehab
* patient moved from an ICU
* GCS≤11 at admission in ICU
* tracheostomy performed for decreased mental status due to the ABI,

Exclusion Criteria:

* tracheostomy performed prior to admission to the ICU
* need for ventilation support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tracheostomy, affected by severe acquired brain injury, hospitalized in our Neurorehabilitation department.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
decannulation time | at data collecting, an average of 1 day
  number days between tracheostomy positioning and removal

SECONDARY OUTCOMES:
length of stay ICU | at data collecting, an average of 1 day
  number days between admission and discharge from ICU
decannulation time in NRiab | at data collecting, an average of 1 day
  number days between NRehab admission and decannulation
Coma Recovery Scale revised score at discharge | at data collecting, an average of 1 day
Glasgow Coma Scale score at discharge | at data collecting, an average of 1 day
Disability Rating Scale Score at discharge | at data collecting, an average of 1 day
Levels of Cognitive Functioning score at discharge | at data collecting, an average of 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona Ed Uniti, CO, Italy